CLINICAL TRIAL: NCT01736293
Title: Natural History of ABCA4-Related Retinopathies
Brief Title: Natural History of Eye Diseases Related to ABCA4 Mutations
Status: Active, not recruiting | Type: Observational
Sponsor: National Eye Institute (NEI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 120203; 12-EI-0203
Record Dates: First submitted 2012-11-27; First posted 2012-11-29 (Estimated); Last update posted 2026-01-28 (Actual); Status verified 2026-01-23

CONDITIONS: Retinal Degeneration; ABCA4-Related Retinopathies
Keywords: Retinal Degeneration; Natural History
MeSH Terms: conditions — Retinal Degeneration

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Affected Participants: Participants with ABCA4-related retinopathies.

SUMMARY:
Background:

- The ABCA4 gene contains a blueprint for the ABCA4 protein. When this protein is absent or faulty (such as in Stargardt s disease), waste material from dead cells collects in the eye. The waste material may cause other cells in the eye to die. This can lead to the loss of vision. Researchers want to look at blood and skin samples from people with ABCA4 gene mutations to study related eye diseases.

Objectives:

- To study eye diseases that are related to mutations in the ABCA4 gene.

Eligibility:

- Individuals at least 12 years of age who have ABCA4 gene mutations.

Design:

* The study requires 12 visits to the National Eye Institute clinic over 10 years. In the first year, there will be three visits. After the first year, participants will have one visit a year for 9 more years.
* Participants will be screened with a physical exam, full eye exam, and medical history. The eye exam will check eye pressure, light and color sensitivity, and retina function.
* Participants will provide a blood sample and a skin tissue sample for study.
* No treatment will be provided as part of this study.

DETAILED DESCRIPTION:
Objectives: The objectives of this study are to 1) establish a cohort of participants with ABCA4-related retinopathies in anticipation of future clinical trials, 2) create a repository of plasma, DNA, and skin fibroblast samples from the accrued cohort of ABCA4-related retinopathy participants, 3) formulate clinical outcome measures for future studies, and 4) acquire and perform preliminary analyses of data that may advance our understanding of genotype-phenotype correlations in ABCA4-related retinopathies.

In addition, the skin fibroblast samples collected from participants may be used to generate iPS cells, which may be differentiated into RPE and/or neural retinal cells. These cells, if produced, will be used to analyze molecular mechanisms involved in disease pathogenesis and to perform high throughput (HTP) drug screens to identify novel potential therapeutic compounds.

Study Population: Sixty-five (65) participants, age 12 or above, with ABCA4-related retinopathies, will be initially accrued for this study. However, up to an additional five participants may be enrolled to replace participants who may withdraw from the study prior to reaching the Month 12 visit.

Design: In this natural history study, participants will be followed for 10 years. Because three years may be required to enroll 65 participants, this study will last up to 13 years. Participants will be recruited through other pre-existing NIH protocols, such as the Ocular Natural History Protocol (16-EI-0134), The Genetics of Inherited Eye Disease Protocol (15-EI-0128), the NEI Screening Protocol (08-EI-0102), and the National Ophthalmic Disease Genotyping and Phenotyping Network, Phase II protocol (eyeGENE II, 10-EI-N164), or through referral from an outside clinician after a review of pertinent medical records and genetic testing. All participants will undergo a standardized medical/ophthalmic history and a complete baseline eye examination, that may include non-invasive electrophysiology (e.g., electroretinography), psychophysiology (e.g., microperimetry, static perimetry), and diagnostic imaging examinations (e.g., optical coherence tomography).

The participants will be examined three times over the course of the first year (i.e., baseline examination, Month 6, and Month 12). After the first year, they will return to the NEI clinic on an annual basis for the next nine years. This study will require a minimum of 12 study visits. Participants may be seen at more frequent intervals at the investigators discretion, depending on the clinical and research situation. Participants will be required to submit a blood sample as part of the study for DNA and serum banking, and they will have the option to provide a 3-mm punch skin biopsy to facilitate research at a cellular level.

Outcome Measures: The primary outcome for this study is the establishment of a cohort of participants with ABCA4-related retinopathies, and the secondary outcome is the creation of a repository of plasma, DNA, and skin fibroblast samples from the accrued cohort of ABCA4-related retinopathy participants. Exploratory outcomes for this study include: 1) the formulation of clinical outcome measures for future studies and 2) the acquisition and preliminary analysis of data that may advance our understanding of genotype-phenotype correlations in ABCA4-related retinopathies. Potential exploratory outcomes include: 1) the generation of iPS cells from the skin fibroblast samples, 2) the differentiation of the generated iPS cells into RPE and/or neural retinal cells, and 3) the use of the participant-specific RPE and/or neural retinal cells to perform HTP drug screens to identify novel potential therapeutic compounds. The cells obtained in this protocol may be genetically modified and may be used for in vivo research.

ELIGIBILITY:
* NCLUSION CRITERIA:

  1. Participant must be 12 years of age or older.
  2. Participant (or legal guardian) must understand and sign the protocol s informed consent document.
  3. Participant must be able to cooperate with detailed psychophysics and electrophysiology testing.
  4. Participant must be able to provide a blood sample.
  5. Participant has:
* A maculopathy or retinal degeneration plus two (or more) clear mutations in the ABCA4 gene (ascertained with CLIA-certified testing) that are known to be associated with retinal disease,

OR

-One clear mutation in ABCA4 associated with a classic presentation of fundus flavimaculatus/Stargardt macular dystrophy (e.g., flecks, macular atrophy) and no pathogenic mutation(s) in other genes known to cause macular dystrophy.

OR

-One clear mutation in ABCA4, a cone-rod degeneration and no clearly pathogenic mutation(s) in other genes known to cause cone-rod degeneration.

EXCLUSION CRITERIA:

Participant has evidence of a systemic condition or ocular disease not related to ABCA4 mutations that would complicate the analysis of psychophysical, electrophysiological, or imaging data. For example, a participant with advanced diabetes mellitus and significant diabetic retinopathy may display changes in retinal function that could be related to either his/her diabetic retinopathy or ABCA4 mutations.

Ages: 12 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Participants will be recruited from other NEI protocols, such as the Ocular Natural History Protocol (16-EI-0134), the Genetics of Inherited Eye Disease Protocol (15-EI-0128), the NEI Screening Protocol (08-EI-0102), and/or the National Ophthalmic Disease Genotyping and Phenotyping Network, Phase II Protocol (eyeGENE II, 10-EI-N164), or through referral from an outside clinician after a review of pertinent medical records and genetic test results.
Sampling Method: Non-Probability Sample
Enrollment: 68 (Actual)
Dates: Start 2012-10-09 (Actual)

PRIMARY OUTCOMES:
Establish cohort | Over the study duration
  Establish a cohort of participants with ABCA4 retinopathies in anticipation of future clinical trials.

CONTACTS AND LOCATIONS:
Overall Officials: Brian P Brooks, M.D., Principal Investigator — National Eye Institute (NEI)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Allikmets R. A photoreceptor cell-specific ATP-binding transporter gene (ABCR) is mutated in recessive Stargardt macular dystrophy. Nat Genet. 1997 Sep;17(1):122. doi: 10.1038/ng0997-122a. No abstract available. PMID 9288113
- [Background] Gomes NL, Greenstein VC, Carlson JN, Tsang SH, Smith RT, Carr RE, Hood DC, Chang S. A comparison of fundus autofluorescence and retinal structure in patients with Stargardt disease. Invest Ophthalmol Vis Sci. 2009 Aug;50(8):3953-9. doi: 10.1167/iovs.08-2657. Epub 2009 Mar 25. PMID 19324865
- [Background] Gonzalez F, Boue S, Izpisua Belmonte JC. Methods for making induced pluripotent stem cells: reprogramming a la carte. Nat Rev Genet. 2011 Apr;12(4):231-42. doi: 10.1038/nrg2937. Epub 2011 Feb 22. PMID 21339765
- [Derived] Pfau M, Huryn LA, Boyle MP, Cukras CA, Zein WM, Turriff A, Ullah E, Hufnagel RB, Jeffrey BG, Brooks BP. Natural History of Visual Dysfunction in ABCA4 Retinopathy and Its Genetic Correlates. Am J Ophthalmol. 2023 Sep;253:224-232. doi: 10.1016/j.ajo.2023.05.014. Epub 2023 May 20. PMID 37211138
- [Derived] Pfau M, Cukras CA, Huryn LA, Zein WM, Ullah E, Boyle MP, Turriff A, Chen MA, Hinduja AS, Siebel HE, Hufnagel RB, Jeffrey BG, Brooks BP. Photoreceptor degeneration in ABCA4-associated retinopathy and its genetic correlates. JCI Insight. 2022 Jan 25;7(2):e155373. doi: 10.1172/jci.insight.155373. PMID 35076026
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2012-EI-0203.html